CLINICAL TRIAL: NCT01476501
Title: Vitamin D Supplementation and Bone Health in Adults With Diabetic Nephropathy
Brief Title: Vitamin D Supplementation in Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, dmager, Associate Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: diabetes vitamin D 20112012
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Sub-optimal Vitamin D Status; Bone Disease; Diabetic Nephropathy
Keywords: vitamin D; bone health; diabetes; nephropathy
MeSH Terms: conditions — Bone Diseases; Diabetic Nephropathies; Diabetes Mellitus; Kidney Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2,000 IU/day vitamin D (Experimental): 2,000 IU/day vitamin D for 6 months (n=60).
  Interventions: Drug: Vitamin D3
- 40,000 IU/month vitamin D (Experimental): 40,000 IU/month for 6 months (n=60).
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Randomized into 1 of 2 oral vitamin D3 softgel capsule supplementation strategies: 1) 2,000 IU/day (2 x 1,000IU/capsule each day) or 2) 40,000 IU/month (4 x 10,000IU/capsule last day of each month), for 6 months each.
  Other Names: Daily: Jamieson NPN 80017530; Monthly: EURO-Pharm DIN 02253178

SUMMARY:
Diabetes is a life-long disease that is getting more common in Canada. One of the most common problems in people with kidney disease is diabetes and low bone mineral density (BMD). This can lead to a higher chance for broken bones, infection and life-long health problems. The most common reason for having low BMD is not getting enough vitamin D (Vit D) in your diet and not having enough sunlight. This is very common in Canada (especially in northern Alberta) because winter is very long. Most people also don't eat or drink enough foods that are high in Vit D (like milk) and so they don't have enough Vit D in their body to make healthy bones. This can mean the only way to get enough Vit D in your body for your bones when you have kidney disease is to take some extra vitamin D in a pill. Most people are not aware that they have poor bone health until they break a bone. Broken bones can really hurt and can prevent a person from being able to walk and take care of themselves. Right now, we are not sure exactly how much Vit D people with diabetes and kidney disease need to take to prevent them from having low BMD or how often they need to take it. Our plan is to study the effect of two ways to take Vit D pills (every day or once a month) on overall Vit D status and on bone health in adult patients with diabetes and chronic kidney disease and see how this influences their quality of life.

Hypotheses:

1. Vitamin D supplementation (2,000 IU/day and 40,000 IU/month) for six months will result in significantly improved overall vitamin D status and improved markers of bone health in adult patients with diabetic nephropathy.
2. Monthly dosing of vitamin D (40,000 IU/month) over six months will result in improved patient adherence and satisfaction with vitamin D supplementation when compared to daily dosing of vitamin D (2000 IU/D). This will improve vitamin D status and bone health parameters, which will result in an increased quality of life and sense of well-being.

DETAILED DESCRIPTION:
Abstract:

Vitamin D has a well-established role in bone health and the prevention of fractures which are associated with increased morbidity and mortality, and reduced quality of life. However, many individuals have sub-optimal vitamin D status (<75nmol/l), and risk increases with geographical location, age, ethnicity, inadequate dietary intake and disease. Diabetes and kidney disease are two chronic diseases associated with both poor bone health and suboptimal vitamin D status. Individuals with diabetes and chronic kidney disease who live in northern Alberta are at a particular risk for suboptimal vitamin D status and poor bone health due to dietary restrictions on vitamin D rich foods (e.g. milk products that are also high in phosphorus and carbohydrates), negligible cutaneous synthesis during the long winter months, and reduced renal capacity to synthesize active vitamin D (1,25(OH)2D). In the general Canadian population, few are able to meet dietary recommendations for vitamin D intake through diet alone and often rely on vitamin D supplements. The need for vitamin D supplementation is increased in diabetics with nephropathy, however the optimal dose and strategy for vitamin D supplementation is unknown. Like other chronic diseases, adherence to therapy is a major issue in this population. With each additional chronic disease an individual has, their adherence to therapy and quality of life decreases. Adherence to vitamin D therapy is known to be particularly poor. This may be related to the silent nature of bone disease, as poor bone health is often not identified until a fracture has occurred. Novel strategies to vitamin D supplementation are needed to prevent poor bone health and fractures, and the resulting decline in quality of life that ensues. Therefore it is important to identify a vitamin D supplementation strategy that increases adherence to vitamin D supplementation and improves vitamin D status and bone health in adults with diabetes and nephropathy.

Objectives:

* Examine the impact of two approaches to oral high dose vitamin D supplementation (2,000 IU/day versus 40,000 IU/month for six months) on overall vitamin D status and markers of bone turnover in adult patients with diabetic nephropathy.
* Examine daily versus monthly vitamin D supplementation strategies in regards to adherence, satisfaction and quality of life in adult patients with diabetic nephropathy.

Hypotheses:

1. Vitamin D supplementation (2,000 IU/day and 40,000 IU/month) for six months will result in significantly improved overall vitamin D status and improved markers of bone health in adult patients with diabetic nephropathy.
2. Monthly dosing of vitamin D (40,000 IU/month) over six months will result in improved patient adherence and satisfaction with vitamin D supplementation when compared to daily dosing of vitamin D (2000 IU/D). This will improve vitamin D status and bone health parameters, which will result in an increased quality of life and sense of well-being.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnoses of diabetes (type 1 or 2) and stage 2-4 chronic kidney disease (glomerular filtration rate: 15-89 ml/min/1.73m2)

Exclusion Criteria:

* Patients with co-morbid conditions known to affect vitamin D metabolism including gastrointestinal, liver, rheumatoid or bone disorders (e.g. hyperthyroidism, untreated celiac disease, cancer, Paget's disease, sarcoidosis, malabsorption, etc). Individuals with severe, permanent vision impairment will be excluded as this will preclude them from reading supplement labels accurately and safely. Pregnant women will be excluded as DXA scans are not recommended during pregnancy. Patients weighing >136kg will be excluded as the DXA table cannot accommodate this weight.
* Patients on drug therapy known to interfere with vitamin D (e.g. oral glucocorticoids, cholestyramine, colestipol, mineral oil, Orlistat, digoxin, antacids).
* Patients with stage 5 CKD (GFR <15ml/min/1.73m2), receiving dialysis or on kidney transplant list.
* Patients with pre-existing hypercalcemia (>2.75mmol/l), hyperphosphatemia (>2.0mmol/l), severe hyperparathyroidism (PTH >600pg/ml), and serum 25(OH)D >200nmol/l.
* Patients with serum 25(OH)D <37.5nmol/l at time of study entry/screening to control for correction of vitamin D deficiency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in serum vitamin D from baseline to 3 and 6 months | Change from baseline to 3 and 6 months
  Changes in serum 25(OH)D and 1,25(OH)D between baseline, 3 and 6 months between individuals and between study arms.

SECONDARY OUTCOMES:
Change in adherence to supplement between 3 and 6 months | 3 and 6 months
  Participant adherence to and acceptance of supplementation strategy will be assessed using a validated questionnaire for adherence in adults with chronic disease.
Change in health related quality of life from baseline to 6 months | baseline and 6 months
  The validated health related quality of life questionnaire SF-36 is often used in renal populations and will be completed at baseline and at 6 months.
Change in dietary intake from baseline to 3 and 6 months | baseline, 3 and 6 months
  3-day food intake records are a validated tool to assess dietary intake, and will consist of 2 weekdays and 1 weekend day. They will be verified by a Registered Dietitian and analyzed using Food Processor (SQL v10 ESHA Research).
Change in 3-day weight-bearing physical activity records from baseline to 3 and 6 months | baseline, 3 and 6 months
  Weight-bearing physical activity will be assessed using a validated questionaire and compared to national recommendations (frequency and duration).
Change in sunlight exposure from baseline to 3 and 6 months | baseline, 3 and 6 months
  A validated sunlight exposure questionnaire will be completed to identify potential for cutaneous vitamin D synthesis based on participants' sun exposure practices.
Change in routine clinical laboratory variables from baseline to 3 and 6 months | baseline, 3 and 6 months
  Routine routine clinical blood work will be assessed for changes following supplementation and for safety. Routine clinical laboratory variables to be collected include: glomerular filtration rate (GFR), urea, creatinine, hemoglobin A1c, fasting blood glucose, albumin, phosphorus, magnesium, and calcium (bound and ionized).
Change in bone health from baseline to 3 and 6 months | Baseline, 3 and 6 months
  Bone mineral density (BMD): Dual-energy x-ray absorptiometry (DXA; gold standard)scan conducted at baseline to characterize bone health.
  Bone turnover markers: Changes in markers of bone formation (osteocalcin and bone specific alkaline phosphatase) and bone resorption (N-telopeptide of type 1 collagen and fibroblast growth factor-23) between baseline and 6 months.
  Serum parathyroid hormone (PTH): Changes in serum PTH will be measured at baseline, 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Diana R Mager, PhD RD, Principal Investigator — University of Alberta; Peter A Senior, MBBS PhD, Principal Investigator — University of Alberta
Locations (1):
- Clinical Research Unit, University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mager DR, Jackson ST, Hoffmann MR, Jindal K, Senior PA. "Vitamin D supplementation and bone health in adults with diabetic nephropathy: the protocol for a randomized controlled trial". BMC Endocr Disord. 2014 Aug 12;14:66. doi: 10.1186/1472-6823-14-66. PMID 25115438
- [Result] Mager DR, Jackson ST, Hoffmann MR, Jindal K, Senior PA. Vitamin D3 supplementation, bone health and quality of life in adults with diabetes and chronic kidney disease: Results of an open label randomized clinical trial. Clin Nutr. 2017 Jun;36(3):686-696. doi: 10.1016/j.clnu.2016.05.012. Epub 2016 Jun 2. PMID 27302208